CLINICAL TRIAL: NCT07065721
Title: CAPAZ-2D: Continuous Glucose Monitoring to Augment and Personalize Self-Management of Type 2 Diabetes in Hispanic/Latinx Young Adults
Brief Title: Continuous Glucose Monitoring for Self-Management of Type 2 Diabetes in Young Adults
Acronym: CAPAZ-2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-8450
Record Dates: First submitted 2025-06-05; First posted 2025-07-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: continuous glucose monitor; type 2 diabetes; young adult
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The intervention consists of a 30-day CGM wear and weekly surveys. Participants will be asked to maintain continuous use of CGM for 30 days and share their CGM data over that period. CGM sensors will be provided free-of-charge. Additionally, participants will be asked to complete weekly electronic surveys measuring self-management behaviors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CGM Wear (Experimental): Participants will wear a continuous glucose monitor for 30 days. They will also wear a FitBit activity tracker watch and complete weekly surveys to report diabetes self-management behaviors.
  Interventions: Device: Continuous glucose monitor

INTERVENTIONS:
Device: Continuous glucose monitor — Participants will wear a continuous glucose monitoring sensor for 30 days. They will also wear a FitBit wrist watch to be able to track their physical activity and they will complete weekly surveys to report diabetes self-management behaviors. After the 30 days, they will participate in a qualitative interview to respond to questions about their experiences.

SUMMARY:
Type 2 diabetes in increasing common in young adults. Utilizing a mixed-methods, community-based approach, this study offers continuous glucose monitors (CGMs) to young adults with type 2 diabetes for 30 days, and collects both quantitative and qualitative data to understand barriers and facilitators of CGM use, participants' changes in awareness of glucose patterns while using the CGM, and preferences for a CGM-based self-management intervention.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes (T2D) is rising in young adults and is associated with increased complications and reduced life expectancy. Poor adherence to diabetes self-management behaviors is common in young adulthood, often leading to poor glycemic control, and existing self-management interventions have had limited effectiveness in this age group. Continuous glucose monitors (CGMs) provide real-time glucose data that can support behavior change and reduce common self-management barriers such as glycemic unawareness, but their use in younger adults is limited. As "digital natives," young adults are well-poised to benefit from CGM interventions, particularly if they reduce barriers of standard self-management education (e.g., time burden). Qualitative data has shown that young adults are interested in CGM use but lack both access to CGMs and understanding of how to best utilize CGM data. The purpose of this proposal is to utilize a mixed-methods, community-engaged approach to generate pilot data for the development of a self-management intervention that pairs CGM glucose data with behavioral data (e.g., FitBit step count, dietary intake) to improve self-management and glycemic awareness and control. Young adults with T2D will be recruited to participate in a 30-day trial wear of CGMs, during which self-management behaviors will also be assessed. Afterward, qualitative interviews with participants will be conducted to understand barriers and facilitators of CGM use, changes in awareness of glucose patterns, and preferences for a CGM-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* adult 18-45 years of age
* diagnosis of type 2 diabetes in the last 5 years, as evidenced in the electronic medical record
* no prior use or experience with wearable CGMs
* possession of a smart phone that is compatible with Dexcom CGM sensors (nearly all smartphones are compatible) and willing to download and utilize the Dexcom CGM app
* fluency in English or Spanish

Exclusion Criteria:

* severe mental illness (e.g., psychosis, suicidal ideation);
* pregnancy or <6 months postpartum

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative data regarding CGM use | Immediately after the intervention
  Semi-structured qualitative interviews will be conducted to understand barriers and facilitators of CGM use, changes in awareness of glucose patterns or relationships between glucose and health behaviors, and preferences for a future CGM-based intervention.

SECONDARY OUTCOMES:
Acceptability and feasibility of CGM wear | Immediately after the intervention
  Mean rating of CGM feasibility, acceptability, utility, satisfaction ≥ 3/5 on a 0-5 scale

OTHER OUTCOMES:
Glucose time-in-range | 30 days (during the intervention period)
  Percent of time that glucose readings are in target range (70-180 mg/dL)
Diabetes self-care behaviors | One week (7 days), last week of the intervention
  Self-report of diabetes self-management behaviors (e.g., healthy eating, physical activity) in the last 7 days using the 13-item Summary of Diabetes Self-care Behaviors Scale (range 0-91, higher = more frequent self-management behaviors).
Diabetes distress | Baseline and follow-up (immediately after the intervention)
  Diabetes distress measured using the Problem Areas in Diabetes scale; range 0-80; higher score = higher diabetes distress
Self-management motivation | Baseline and follow-up (immediately after the intervention)
  Motivation and attitudes about behavioral diabetes self-management utilizing the 9-item Motivation and Attitudes Toward Changing Health measure (range: 9-45, higher scores = greater motivation/more positive attitude).
Self-reported physical activity | Baseline and follow-up (immediately after the intervention)
  Self-reported moderate and vigorous physical activity using the International Physical Activity Questionnaire (scored as metabolic equivalent units per week)
Objectively measured physical activity | 30 days (during the intervention period)
  FitBit-sensed step count (weekly average)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L McCurley, PhD MPH, Principal Investigator — San Diego State University
Locations (1):
- Scripps Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to the very small size of this study, data will not be shared, as there is risk of identifying participants.